CLINICAL TRIAL: NCT05452590
Title: Wire-in-needle vs. Traditional Technique for Ultrasound-guided Central Venous Catheter Placement - a Randomized Controlled Trial (The WIN-Study)
Brief Title: Wire-in-needle vs. Traditional Technique for Ultrasound-guided Central Venous Catheter Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Kristen Thomsen, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-100852-BO-ff
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Central Venous Catheter Placement
MeSH Terms: interventions — Central Venous Catheters

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided wire-in-needle technique (Experimental): The guidewire will be connected to the needle. The IJV will be punctured in a long-axis in-plane approach. When the needle tip enters the IJV, the guidewire will be advanced through the needle into the IJV under continuous ultrasound visualization. The needle will then be removed. The correct guidewire position in the IJV will be confirmed in the long-axis and short-axis view. Afterwards, the second guidewire will be placed in the same IJV approximately 1-2 centimeters distal to the fist guidewire using the same technique. The correct guidewire position in the IJV will be confirmed in the long-axis and short-axis view again.
  Interventions: Procedure: Ultrasound-guided wire-in-needle technique for central venous catheter placement
- Traditional technique (No Intervention): A syringe will be connected to the needle. The IJV will be punctured in a long-axis in-plane or short-axis out-of-plane approach (as preferred by the anesthesiologist). When the needle tip enters the IJV, blood is aspirated using the syringe. The operator will then discontinue US-guidance, disconnect the syringe and advance the guidewire through the needle into the IJV. The needle will then be removed. The correct guidewire position in the IJV will be confirmed in the long-axis and short-axis view. Afterwards, the second guidewire will be placed in the same IJV approximately 1-2 centimeters distal to the fist guidewire using the same technique. The correct guidewire position in the IJV will be confirmed in the long-axis and short-axis view again.

INTERVENTIONS:
Procedure: Ultrasound-guided wire-in-needle technique for central venous catheter placement — The guidewire will be connected to the needle. The IJV will be punctured in a long-axis in-plane approach. When the needle tip enters the IJV, the guidewire will be advanced through the needle into the IJV under continuous ultrasound visualization. The needle will then be removed. The correct guidewire position in the IJV will be confirmed in the long-axis and short-axis view. Afterwards, the second guidewire will be placed in the same IJV approximately 1-2 centimeters distal to the fist guidewire using the same technique. The correct guidewire position in the IJV will be confirmed in the long-axis and short-axis view again.
  Arms: Ultrasound-guided wire-in-needle technique

SUMMARY:
Central venous catheters (CVC) are commonly inserted in surgical or critically ill patients. However, CVC placement can cause severe complications. To reduce the incidence of complications and increase procedural safety and quality, ultrasound (US)-guided CVC insertion is recommended by various scientific societies, including the American Society of Anesthesiologists.

During conventional US-guided CVC placement, the correct position of the needle tip in the venous vessel is confirmed by direct US visualization and aspiration of blood using a syringe connected to the needle. After blood aspiration, the operator must discontinue US-guidance to disconnect the syringe and the needle and to pass the guidewire through the needle (without direct US visualization). This step bears the risks of dislocating the needle tip and puncturing the posterior wall of the target vein or an adjacent artery.

Some authors thus propose an US-guided wire-in-needle technique - in which the guidewire is directly adapted to the needle (without a syringe) from the beginning of the procedure and the guidewire is advanced under direct US visualization. Whether the wire-in-needle technique decreases the procedure time, the number of needle passes, and complications compared to conventional US-guided CVC remains scarcely investigated. We thus propose a randomized controlled trial to investigate whether the US-guided wire-in-needle technique for CVC placement in the internal jugular vein (IJV) is faster and safer than the conventional US-guided technique in patients having cardiac surgery.

DETAILED DESCRIPTION:
Patients scheduled for elective cardiac surgery receive a CVC and sheath introducer central line in the same internal jugular vein. Both catheters require the insertion of a guidewire into the vein to insert the catheter (seldinger technique). The anesthesiologist is going to place both guidewires before advancing the catheters over the guidewires.

The IJV will be examined before catheter placement to confirm that a long-axis view is possible. The right IJV will be chosen for CVC and sheath introducer central line placement. Patients will be then randomized to the US-guided wire-in-needle technique or the conventional US-guided technique just before catheter placement. Randomization will thus be concealed until the last practical moment. The patients will be randomized by a computer algorithm. Patients will be blinded to group allocation.

Anesthesiologists inserting the catheters will have at least 2-month experience in both US-guided wire-in-needle technique or the conventional US-guided technique. Patients will be equipped with basic anesthetic monitoring (electrocardiogram, pulse oximetry, upper-arm cuff oscillometry) and an arterial catheter. All patients will be intubated and mechanically ventilated during the procedure. The patient will be placed in a 15° Trendelenburg position. Catheter placement will be performed under sterile conditions with the US probe covered with a sterile cover.

US-guided wire-in-needle technique The guidewire will be connected to the needle. The IJV will be punctured in a long-axis in-plane approach. When the needle tip enters the IJV, the guidewire will be advanced through the needle into the IJV under continuous ultrasound visualization. The needle will then be removed. The correct guidewire position in the IJV will be confirmed in the long-axis and short-axis view. Afterwards, the second guidewire will be placed in the same IJV approximately 1-2 centimeters distal to the fist guidewire using the same technique. The correct guidewire position in the IJV will be confirmed in the long-axis and short-axis view again.

Traditional technique A syringe will be connected to the needle. The IJV will be punctured in a long-axis in-plane or short-axis out-of-plane approach (as preferred by the anesthesiologist). When the needle tip enters the IJV, blood is aspirated using the syringe. The operator will then discontinue US-guidance, disconnect the syringe and advance the guidewire through the needle into the IJV. The needle will then be removed. The correct guidewire position in the IJV will be confirmed in the long-axis and short-axis view. Afterwards, the second guidewire will be placed in the same IJV approximately 1-2 centimeters distal to the fist guidewire using the same technique. The correct guidewire position in the IJV will be confirmed in the long-axis and short-axis view again.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective cardiac surgery at the University Heart Center Hamburg-Eppendorf in whom CVC placement and sheath introducer central line placement in the internal jugular vein is indicated for clinical reasons unrelated to the study
* age > 18 years
* Written informed consent

Exclusion Criteria:

* longitudinal (long axis) view cannot be performed because of anatomical reasons (e.g., short neck).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Time between skin puncture and removal of the needle during placement of the first guidewire. | From the beginning of central venous catheter placement till the end of central venous catheter placement.
  Time between skin puncture and removal of the needle during placement of the first guidewire in seconds.

SECONDARY OUTCOMES:
Complications | From the beginning of central venous catheter placement till the end of central venous catheter placement.
  arterial puncture
Complications | From the beginning of central venous catheter placement till the end of central venous catheter placement.
  posterior wall puncture/hematoma
Complications | From the beginning of central venous catheter placement till the end of central venous catheter placement.
  cervical hematoma
Number of needle passes | From the beginning of central venous catheter placement till the end of central venous catheter placement.
  Number of needle passes required to place the wire in the vessel
Number of skin punctures | From the beginning of central venous catheter placement till the end of central venous catheter placement.
  Number of skin punctures required to place the wire in the vessel
First-pass success rate | From the beginning of central venous catheter placement till the end of central venous catheter placement.
  First-pass success rate for placing the wire in the vessel

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No